CLINICAL TRIAL: NCT01206452
Title: Use of Oral Steroids Before Circumferential Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation to Improve Outcomes
Brief Title: Oral Steroids Before Pulmonary Vein Isolation to Improve Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12153
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation plus prednisone (Experimental): Participants undergo ablation procedure and receive predinisone at protocol determined times.
  Interventions: Drug: Prednisone; Procedure: Ablation Procedure
- Ablation plus placebo (Placebo Comparator): Participants undergo ablation procedure and receive placebo at protocol determined times.
  Interventions: Other: Placebo; Procedure: Ablation Procedure

INTERVENTIONS:
Drug: Prednisone — 60mg of oral prednisone 2 days before procedure, day of procedure, and 1 day after procedure
  Arms: Ablation plus prednisone
Other: Placebo — 60mg placebo pill given 2 days before procedure, day of procedure, and 1 day after procedure
  Arms: Ablation plus placebo
Procedure: Ablation Procedure — Atrial Fibrillation (AF) ablation

SUMMARY:
The primary purpose of this study is to assess the efficacy of oral prednisone in improving the outcomes of pulmonary vein isolation with radiofrequency ablation.

DETAILED DESCRIPTION:
The purpose of this study is:

1. To assess the efficacy of oral prednisone in improving the outcomes of pulmonary vein isolation with radiofrequency ablation.
2. To measure the inflammatory cytokine (TNF-α, IL-1, IL-6, IL-8) response to radiofrequency ablation for atrial fibrillation with or without prior prednisone treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent;
2. Scheduled for radiofrequency ablation procedure for treatment of atrial fibrillation

Exclusion Criteria:

1. History of heart failure (right or left or biventricular) or cardiomyopathy.
2. Immunosuppressive disorders and systemic fungal infection
3. Concurrent use of corticosteroids in one week prior recruitment.
4. Allergy or prednisone or its components.
5. Other medical conditions were use of corticosteroids is not recommended or contraindicated.
6. Patients with chronic and permanent atrial fibrillation.
7. Patients with established diagnosis of rheumatological and immunological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.23 (8.95) | 63 (8.69) | 63.12 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 22 | 24 | 46
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.48 (5.19) | 30.53 (5.93) | 29.51 (5.63)
AF Duration [Mean (Standard Deviation); unit: years] | 7.92 (7.66) | 4.98 (4.81) | 6.45 (6.45)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Atrial Fibrillation Recurrence From 6 Months up to 12 Months
Description: Number of AF recurrences between the two study groups as assessed by 1-month event monitor placed at 6 and 12 months post-ablation. Any episode of AF lasting greater than 30 seconds was counted as a recurrence.
Time Frame: From 6 months up to 12 months post-procedure
Measure: Number; unit: Participants with AF recurrence
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Number analyzed (Participants) | 30 | 30
Participants with AF recurrence | 4 | 6

2. Secondary Outcome: Number of Participants With Atrial Fibrillation Recurrence From 0 Months up to 3 Months
Description: Number of AF recurrences between the two study groups as assessed by inpatient telemetry in the immediate post-procedure period until discharge and 1-month event monitor placed at 3 months post-ablation. Any episode of AF lasting greater than 30 seconds was counted as a recurrence.
Time Frame: From 0 months up to 3 months post procedure
Measure: Number; unit: Participants with AF recurrence
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Number analyzed (Participants) | 30 | 30
Participants with AF recurrence | 6 | 8

3. Secondary Outcome: Number of Participants With Atrial Fibrillation Recurrence From 3 Months up to 6 Months
Description: Number of AF recurrences between the two study groups as assessed by 1-month event monitor placed at 3 and 6 months post-ablation. Any episode of AF lasting greater than 30 seconds was counted as a recurrence.
Time Frame: From 3 months up to 6 months post-procedure
Measure: Number; unit: Participants with AF recurrence
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Number analyzed (Participants) | 30 | 30
Participants with AF recurrence | 5 | 9

4. Secondary Outcome: Inflammatory Cytokine Response to Ablation Procedure
Description: Measure inflammatory marker levels, including IL-1, IL-6, IL-8, and TNF-α, immediately post-ablation in keeping with prior studies on the anti-inflammatory effects of steroids following cardiac surgery.
Time Frame: Immediately Post-Ablation Procedure
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Number analyzed (Participants) | 30 | 30
pg/ml
  IL-1 level | 11 (2.8) | 7.94 (2.1)
  IL-8 level | 15.3 (8.14) | 10.54 (9.63)
  TNF-α level | 7.9 (3.2) | 5.45 (2.6)
  IL-6 level | 15.78 (13.19) | 9.03 (7.026)

5. Secondary Outcome: Inflammatory Cytokine Response to Ablation Procedure
Description: Measure inflammatory marker levels, including IL-1, IL-6, IL-8, and TNF-α, 24 hours post-ablation to assess interval response to steroid administration.
Time Frame: 24 Hours after Ablation Procedure
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Number analyzed (Participants) | 30 | 30
pg/ml
  IL-1 level | 11.7 (15.4) | 8.5 (12.1)
  IL-8 level | 59.6 (54.9) | 63.9 (52.8)
  TNF-α level | 9.7 (15.8) | 7.5 (16.1)
  IL-6 level | 40.9 (39.9) | 40.2 (49.7)

ADVERSE EVENTS:
Arm/Group | Ablation Plus Placebo | Ablation Plus Prednisone
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Plus Placebo (N=30) | Ablation Plus Prednisone (N=30)
Groin hematoma (Blood and lymphatic system disorders) | 3 (3) | 2 (2) — Related to ablation procedure. No subjects required blood transfusions or surgical repair.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes